CLINICAL TRIAL: NCT05548205
Title: Effect of 2-Week Continuous Glucose Monitoring on Glycemic Management in Patients New-to-Insulin on Hospital Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01051
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Diabetes
Keywords: Continuous Glucose Monitoring (CGM)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Continuous Glucose Monitoring (CGM) (Experimental): Patients in the CGM group will be instructed to wear a CGM uninterruptedly for 2 weeks duration.
  Interventions: Device: Continuous Glucose Monitor
- Blood Glucose Monitoring (BGM) (Active Comparator): Patients in the BGM group will be instructed to check their blood glucose utilizing fingerstick glucose monitoring multiple times daily depending on their insulin regimen for 2 weeks duration.
  Interventions: Device: Blood Glucose Monitor

INTERVENTIONS:
Device: Continuous Glucose Monitor — Manufactured by Abbott Diabetes Care Inc. Administered by trained investigator prior to hospital discharge, left in place for 2 weeks duration, then removed.
  Other Names: Dexcom G7
  Arms: Continuous Glucose Monitoring (CGM)
Device: Blood Glucose Monitor — Self-administered according to investigator instruction.
  Arms: Blood Glucose Monitoring (BGM)

SUMMARY:
The proposed study will be a randomized, prospective, non-blinded study of 120 participants with type 1 or type 2 diabetes that are new-to-insulin on hospital discharge. On hospital discharge, participants will be assigned to either the intervention of wearing a continuous glucose monitor (CGM) for 2 weeks or blood glucose monitoring (BGM) for 2 weeks. They will have a 2-week follow up visit, during which insulin doses will be adjusted as needed, and a 3-month follow-up visit, at which point HbA1c will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-100 years
2. Known history of type 1 or type 2 diabetes
3. Admitted to NYU Langone Hospital - Long Island between December 16, 2024- December 31, 2026
4. New initiation of insulin therapy, including basal insulin regimen, basal-bolus insulin regimen, or mixed insulin regimen at the time of hospital discharge

Exclusion Criteria:

1. Prior to admission use of home insulin therapy
2. Current use of systemic corticosteroids
3. Active pregnancy; as pregnancy requires different blood glucose targets, subjects known to be pregnant will be excluded from this study. Subjects will not be tested for pregnancy outside of testing performed in routine medical care; pregnancy will be determined by patient self-reporting. Females of childbearing potential will not be instructed to avoid pregnancy, however if they became pregnant during the study (detected by self-reporting), they will be withdrawn from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Hemoglobin A1c (HbA1c) | Baseline, Month 3 Post-Discharge
  Assessed via CGM or BGM.

SECONDARY OUTCOMES:
Number of Hospital Admissions | Up to Month 3 Post-Discharge
Number of Emergency Department (ER) Visits | Up to Month 3 Post-Discharge
Number of Hypoglycemic Events | Up to Month 3 Post-Discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldstein, Principal Investigator — NYU Langone Hospital - Long Island
Locations (1):
- NYU Langone Hospital - Long Island, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Stanislaw Klek (Stanislaw.Klek@nyulangone.org). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to Stanislaw.Klek@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.